CLINICAL TRIAL: NCT03342521
Title: Optical Frequency Domain Imaging-Quantified Intracoronary Thrombus Mass During Primary Percutaneous Coronary Intervention, Its Relationship With Antiplatelet Pretreatment Effect And Its Impact On Myocardial Reperfusion
Brief Title: OFDI-Quantified Intracoronary Thrombus, Antiplatelet Pretreatment Effect and Myocardial Reperfusion
Acronym: ODIPP
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 17-107
Record Dates: First submitted 2017-10-19; First posted 2017-11-17 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2017-11

CONDITIONS: Myocardial Infarction; Thrombosis, Coronary
Keywords: myocardial infarction; optical coherence tomography; intracoronary thrombus; VerifyNow
MeSH Terms: conditions — Myocardial Infarction; Coronary Thrombosis | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: optical coherence tomography and VerifyNow — optical coherence tomography Imaging P2Y12 and Aspirin reaction units quantification by the VerifyNow

SUMMARY:
The management of ST-elevation myocardial infarction in the acute phase requires an optimal antiaggregation combining aspirin and a P2Y12 inhibitor (clopidogrel, prasugrel or ticagrelor). Primary percutaneous coronary intervention must be performed within 2 hours of first medical contact. However, even with the new P2Y12 inhibitors, effective platelet inhibition which is required to inhibit the progression of intracoronary thrombus, is present only in half of the patients at 2 hours.

Optical coherence tomography (OCT) is the reference method for visualizing and quantifying intracoronary thrombus. The post-stenting intracoronary residual mass evaluated in OCT was associated with altered myocardial reperfusion indices, which were themselves associated with the prognosis of the patient. However, the determinants of this post-stenting residual mass -mostly thrombotic- remain unknown.

Measurement of platelet reactivity (expressed as P2Y12 Reaction Unit and Aspirin Reaction Unit) by simple turbidimetric tests (VerifyNow) is available in the cathlab. Enhanced platelet reactivity is reported in patients with acute coronary syndrome and represents a high-risk situation for recurrent coronary events in this setting.

The study aims to:

1. to evaluate the relationship between the post-stenting residual intracoronary mass evaluated in OCT and the platelet response at the time of the PCI evaluated by Verify Now
2. to confirm the impact of the residual mass measured by OCT on the EKG and angiographic myocardial reperfusion indices
3. identify patients with high thrombotic risk who may require more intensive antithrombotic therapy
4. identify simple biological markers associated with the residual mass measured by OCT

ELIGIBILITY:
Inclusion Criteria:

* primary PCI with successful stenting for ST-elevation myocardial infarction
* pretreated with ticagrelor, aspirin and enoxaparin
* OCT and verifyNow performed in the acute phase

Exclusion Criteria:

* stent thrombosis
* known coagulation disorder
* clinical instability
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted in our hospital for primary PCI for ST-elevation myocardial infarction treated with successful stenting who had OCT and VerifyNow in the acute phase
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
the volume of residual intrastent mass measured by OCT | day 0
  volume of the residual mass in mm3
the platelet reactivity assessed by VerifyNow | day 0
  P2Y12 and aspirin reaction units, assessed by VerifyNow

SECONDARY OUTCOMES:
regression of EKG ST-segment elevation | day 0
  regression of ST-segment elevation >50% after angioplasty
Corrected Timi Frame count | day 0
  TIMI frame count (number) assessed after angioplasty
Myocardial blush grade | day 0
  Blush grade (from 0= no blush; 1=minimal; 2=moderate to 3= normal blush) assessed on angiography after angioplasty
angiographic pre-stenting thrombus grade | day 0
  angiographic thrombus grade score (from 0=no thrombus to 5=occlusive thrombus)
troponin | day 0
  biological marker (µg/L)
fibrinogen | day 0
  biological marker (in g/L)
albumin | day 0
  biological marker (in g/L)

CONTACTS AND LOCATIONS:
Overall Officials: vincent ROULE, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- CAEN University Hospital, Caen, France